CLINICAL TRIAL: NCT06394401
Title: Optimized Carbohydrate Fueling to Enhance Physical Performance During Energy Deficit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-15H
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Energy Supply; Deficiency

STUDY DESIGN:
Intervention Model Description: Double blinded randomized crossover design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Energy Balance: Glucose (Active Comparator): Following 48 hours of consuming an energy balance diet, volunteers complete 80 min of steady-state (60 ± 5% V̇O2peak) exercise on a cycle ergometer while consuming 80 g of glucose
  Interventions: Dietary Supplement: BAL:GLU
- Energy Balance: Glucose plus Fructose (Experimental): Following 48 hours of consuming an energy balance diet, volunteers complete 80 min of steady-state (60 ± 5% V̇O2peak) exercise on a cycle ergometer while consuming 53 g of glucose and 27 g of fructose.
  Interventions: Dietary Supplement: BAL:GLU+FRU
- Energy Deficit: Glucose (Active Comparator): Following 48 hours of consuming an energy deficit diet, volunteers complete 80 min of steady-state (60 ± 5% V̇O2peak) exercise on a cycle ergometer while consuming 80 g of glucose
  Interventions: Dietary Supplement: DEF:GLU
- Energy Deficit: Glucose plus Fructose (Experimental): Following 48 hours of consuming an energy deficit diet, volunteers complete 80 min of steady-state (60 ± 5% V̇O2peak) exercise on a cycle ergometer while consuming 53 g of glucose and 27 g of fructose.
  Interventions: Dietary Supplement: DEF:GLU+FRU

INTERVENTIONS:
Dietary Supplement: BAL:GLU — 80 g glucose consumed during steady-state exercise following 48 hours of consuming an energy balance diet
  Arms: Energy Balance: Glucose
Dietary Supplement: BAL:GLU+FRU — 53 g glucose plus 27 g fructose consumed during steady-state exercise following 48 hours of consuming an energy balance diet
  Arms: Energy Balance: Glucose plus Fructose
Dietary Supplement: DEF:GLU — 80 g glucose consumed during steady-state exercise following 48 hours of consuming an energy balance diet
  Arms: Energy Deficit: Glucose
Dietary Supplement: DEF:GLU+FRU — 53 g glucose plus 27 g fructose consumed during steady-state exercise following 48 hours of consuming an energy balance diet
  Arms: Energy Deficit: Glucose plus Fructose

SUMMARY:
This randomized crossover study will examine the effects of consuming isocaloric GLU+FRU or GLU alone on rates of exogenous carbohydrate oxidation during aerobic exercise and physical performance (time trial) under energy balance (BAL) and energy deficit (DEF). Baseline data will be collected on volunteer height, weight, body composition, and V̇O2peak. To ensure volunteers are familiar with exercise protocols, they will complete practice sessions of all exercise before the start of data collection. Exercise and diet will be controlled throughout data collection. To start the protocol volunteers will complete a bout of glycogen normalization on a cycle ergometer followed by 48 hours of refeeding at 100% (BAL) or 50% (DEF) of their energy needs. After the 48 hours of refeeding volunteers will return to the laboratory to complete 80 min of steady-state (60 ± 5% V̇O2peak) exercise on a cycle ergometer. Immediately before and during steady-state exercise, volunteers will consume either 80 g of GLU+FRU (53 g glucose + 27 g fructose) or 80 g GLU. Drinks containing corn-derived crystalline fructose (KRYSTAR® 300, Tate and Lyle Sugars, London, UK) and glucose (CERELOSE®, Ingredion, Westchester, IL, USA) will be prepared by unblinded USARIEM staff. Drinks will be enriched with 13C stable isotopes (Cambridge Isotope Laboratory, Andover, MA, USA) to measure exogenous and plasma carbohydrate oxidation during steady-state exercise. After steady-state exercise, physical performance will be assessed using a graded exercise test on a stationary bike. Indirect calorimetry and breath sampling will be used to determine substrate oxidation during steady-state exercise. Serial blood draws will be collected during each trial to assess isotope enrichments, and circulating substrate/hormone responses. Muscle biopsies will be performed before and after steady-state exercise to assess glycogen status, enzyme activity, and molecular regulation of substrate metabolism. There will be a minimum of 7 days between each carbohydrate metabolism study day.

DETAILED DESCRIPTION:
Periods of energy deficit (DEF) contribute to declines in physical performance during military operations. During DEF, glucose (GLU) supplementation alone is likely an insufficient intervention to enhance physical performance. The lack of an ergogenic effect with GLU consumption during DEF may result from lower glucose uptake and exogenous glucose oxidation in peripheral tissue. As the current carbohydrate beverage base in Meals, Ready-to-Eat (MRE) is derived solely from GLU, an alternative ration product may be needed to enhance physical performance during DEF. Use of multiple transportable carbohydrates, such as glucose plus fructose (GLU+FRU) may be a more effective ration product, as it has been shown to increase rates of exogenous carbohydrate oxidation and improve physical performance compared to GLU. However, previous studies have only been conducted during energy balance (BAL), and the influence of GLU+FRU on substrate oxidation and physical performance compared to GLU during DEF is currently unknown. This randomized crossover placebo controlled double blinded study will examine the effects of consuming GLU compared to GLU+FRU on substrate oxidation and physical performance during metabolically-matched, steady-state exercise during BAL and DEF. Twelve healthy, recreationally active men and women between the ages of 18-39 yrs will be required to complete this study. To start the protocol volunteers will complete a bout of glycogen normalization cycling followed by 48 hours of refeeding at 100% (BAL) or 50% (DEF) of their energy needs. After the 48 hours refeeding volunteers will return to the laboratory and complete 80 min of steady-state (60 ± 5% VO2peak) cycling. Immediately before and during steady-state exercise, volunteers will consume either 80 g of GLU+FRU (53 g glucose + 27 g fructose) or 80 g GLU. Drinks will be enriched with 13C stable isotopes to measure exogenous carbohydrate oxidation during steady-state exercise. After steady-state exercise, aerobic performance will be assessed. Indirect calorimetry and breath sampling will be used to determine substrate oxidation during steady-state exercise. Serial blood draws will be collected during each trial to assess isotope enrichments, and circulating substrate/hormone responses. Muscle biopsies will be performed before and after steady-state exercise to assess glycogen status, enzyme activity, and molecular regulation of substrate metabolism. Volunteers will complete all four trials (BAL: GLU, DEF: GLU, BAL: GLU+FRU, DEF: GLU+FRU) in a randomized order under controlled laboratory conditions at USARIEM. There will be a minimum of 7 days between each carbohydrate metabolism study day.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 39 years
* Healthy without evidence of chronic illness or musculoskeletal injury as determined by the USARIEM Office of Medical Support and Oversight (OMSO) or home duty station medical support
* Routinely participate in aerobic and/or resistance exercise at least 2 days per week
* Willing to refrain from alcohol, smoking/using any nicotine product (includes e-cigarettes, vaping, chewing tobacco), caffeine, and dietary supplements while consuming the study diet
* Supervisor approval for federal civilian employees and non-HRV active duty military personnel
* Females must have normal menstrual cycles between 26-32 days in duration; 5 menstrual cycles within the past 6 months; or on continuous oral or IUD contraception without placebo.

Exclusion Criteria:

* Musculoskeletal injuries that compromise exercise capability
* Metabolic or cardiovascular abnormalities, gastrointestinal disorders (e.g., kidney disease, diabetes, cardiovascular disease, etc.), claustrophobia
* Significantly abnormal blood clotting as determined by OMSO or home duty station medical support
* Allergy to lidocaine (or similar local anesthetic)
* Present condition of alcoholism, anabolic steroid use, or other substance abuse issues as determined by OMSO or home duty station medical support
* Blood donation within 8-wk of beginning the study
* Pregnant, trying to become pregnant, and/or breastfeeding (results of urine pregnancy test and self-report for breastfeeding will be obtained before body composition testing)
* Unwilling or unable to consume study diets or foods provided due to personal preference, dietary restrictions, and/or food allergies
* Unwilling or unable to adhere to study physical restrictions

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Exogenous carbohydrate oxidation | 80 minutes
  Determine the effects of consuming glucose compared to glucose plus fructose on the rate (g/min) of exogenous carbohydrate oxidation during metabolically-matched steady-state exercise during energy balance and deficit.

SECONDARY OUTCOMES:
Time to exhaustion | 20 minutes
  Determine the effects of consuming glucose compared to glucose plus fructose on time to exhaustion (min) during a graded exercise performance test during energy balance and deficit.

CONTACTS AND LOCATIONS:
Locations (1):
- USARIEM, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No